CLINICAL TRIAL: NCT01272375
Title: An Open Study To Estimate The Plasma Pharmacokinetics Of PF-04764793 Administered Via Oral Inhalation Using Dry Powder Inhalers
Brief Title: This Study Is To Estimate The Time Course Of Pf-04764793 In The Blood Following Dosing By Oral Inhalation From Dry Powder Inhalers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1691011
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Treatment A PF-04764793 (Experimental): PF-04764793 using inhaler A
  Interventions: Drug: Treatment A
- Treatment B PF-04764793 (Experimental): PF-04764793 using inhaler A
  Interventions: Drug: Treatment B
- Treatment C PF-04764793 (Experimental): PF-04764793 using inhaler A
  Interventions: Drug: Treatment C
- Treatment D PF-04764793 (Experimental): PF-04764793 using inhaler A
  Interventions: Drug: Treatment D
- Treatment E PF-04764793 (Experimental): PF-04764793 using inhaler B
  Interventions: Drug: Treatment E
- Treatment F PF-04764793 (Experimental): PF-04764793 using inhaler B
  Interventions: Drug: Treatment F
- Treatment G PF-04764793 (Experimental): PF-04764793 using inhaler B
  Interventions: Drug: Treatment G

INTERVENTIONS:
Drug: Treatment A — PF-04764793 250/50 using inhaler A
  Arms: Treatment A PF-04764793
Drug: Treatment B — PF-04764793 250/50 using inhaler A
  Arms: Treatment B PF-04764793
Drug: Treatment C — PF-04764793 250/50 using inhaler A
  Arms: Treatment C PF-04764793
Drug: Treatment D — PF-04764793 250/50 using inhaler A
  Arms: Treatment D PF-04764793
Drug: Treatment E — PF-04764793 250/50 using inhaler B
  Arms: Treatment E PF-04764793
Drug: Treatment F — PF-04764793 250/50 using inhaler B
  Arms: Treatment F PF-04764793
Drug: Treatment G — PF-04764793 250/50 using inhaler B
  Arms: Treatment G PF-04764793

SUMMARY:
The purpose of this study is to investigate the time course of PF-04764793 concentration in the blood following dosing by oral inhalation from dry powder inhalers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m^2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 14 drinks/week for females or 21 drinks/week for males.
* Pregnant or nursing females.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameter: Area under the curve (AUClast)from the time of dosing to the last data point taken for PF-04764793 | 48 hours
Plasma pharmacokinetic parameter: Maximum concentration (Cmax) for PF-04764793 in plasma. | 48 hours

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameter: Area under the curve (AUC0-24) from time of dosing to 24 hours post dose for PF-04764793. | 48 hours
Plasma pharmacokinetic parameter: Area under the curve (AUCinf) from the time of dosing extrapolated to infinity for PF-04764793. | 48 hours
Plasma pharmacokinetic parameter: Time of maximum (Tmax) concentration of PF-04764793 in plasma. | 48 hours
Plasma pharmacokinetic parameter: Terminal half-life of PF-04764793. | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1691011&StudyName=An%20Open%20Study%20To%20Estimate%20The%20Plasma%20Pharmacokinetics%20Of%20PF-04764793%20Administered%20Via%20Oral%20Inhalation%20Using%20Dry%20Powder%20Inhalers